CLINICAL TRIAL: NCT06080191
Title: Phase I Clinical Trial on the Use of Fresh, Allogeneic, Second-generation CD19-CAR T Cells for Treatment of Children With Relapsed/Refractory B-cell Acute Lymphoblastic Leukemia
Brief Title: Allogeneic Second-generation CD19-CAR T Cells for Pediatric Relapsed/Refractory B-ALL
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Bambino Gesù Hospital and Research Institute (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: AlloCAR
Record Dates: First submitted 2023-09-12; First posted 2023-10-12 (Actual); Last update posted 2025-12-02 (Actual); Status verified 2025-11

CONDITIONS: B-cell Acute Lymphoblastic Leukemia
Keywords: B-cell acute lymphoblastic leukemia; Children; Adolescent; Young adults
MeSH Terms: conditions — Burkitt Lymphoma

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Single arm (Experimental): A single IV infusion of CD19-CAR_Lenti_ALLO (allogeneic CD19-directed chimeric antigen receptor T-cells) on Day 0 after lymphodepletion. Patients will be divided in two cohorts based on donor HLA matching: cohort A (fully matched, familial or unrelated donor); cohort B (haploidentical donor).
  Patients will receive the following lymphodepletion:
  * Fludarabine (Flu) 30 mg/m2 per day on days -5, -4 and -3
  * Cyclophosphamide (Cyclo) 1000 mg/m2 per day on days -5, -4 and -3.
  CD19-CAR_Lenti_ALLO will be infused at the following dose levels:
  Cohort A:
  * DL1: 3.0 x10^6 CAR+ cells/kg
  * DL2: 5.0x10^6 CAR+ cells/kg
  Cohort B:
  * DL1: 1x10^6 CAR+ cells/kg
  * DL2: 3x10^6 CAR + cells/kg
  If 2 DLT are observed in the dose level 1, an additional DL0 of 2.0x10^6 CAR+ cells/kg (cohort A) or 0.5x10^6 CAR+ cells/kg (cohort B) will be explored.
  Interventions: Drug: CD19-CAR_Lenti_ALLO

INTERVENTIONS:
Drug: CD19-CAR_Lenti_ALLO — Biological/Vaccine: CD19-CAR_Lenti_ALLO
  A single infusion of CD19-CAR_Lenti_ALLO on Day 0

SUMMARY:
This is a phase I, open label study to evaluate the safety, identify the recommended dose (RD) and obtain preliminar evidence of the efficacy of allogeneic, CD19-directed Chimeric Antigen Receptor T (alloCAR-T) cells in pediatric and young adults patients with relapsed/refractory B-cell precursor Acute Lymphoblastic Leukemia (BCP-ALL).

DETAILED DESCRIPTION:
This is a phase 1, single-center, non-randomized, open-label, dose-escalation study to evaluate the safety, identify the recommended dose (RD) and obtain preliminar evidence of the efficacy of fresh, donor-derived, CD19-directed-second-generation CAR T cells (alloCART) in pediatric and young adults patients with relapsed/refractory B-cell precursor Acute Lymphoblastic Leukemia (BCP-ALL) occurring either after allogeneic hematopoietic stem cell transplantation (alloHSCT) or before alloHSCT, in case of refractory disease and availability of a HLA-fully matched donor.

ELIGIBILITY:
Patient Inclusion Criteria:

1. Patients with a diagnosis of CD19 expressing B ALL relapse, and one of the following:

   1. Relapse after alloHSCT OR
   2. Relapsed/refractory disease, with failure of frontline therapy and at least 2 rescue strategies, including CD19/CD22-directed monoclonal antibody and availability of a fully matched related donor.
2. CD19+ count ≥ 50 cells/mcl and/or Minimal Residual Disease (MRD) ≥ 10^-4.
3. Voluntary informed consent. For subjects < 18-years old their legal guardian must give informed consent. Pediatric subjects will be included in age-appropriate discussion and verbal assent will be obtained for those greater than or equal to 12 years of age, when appropriate.
4. Clinical performance status: patients > 16 years of age: Karnofsky greater than or equal to 60%; patients ≤ 16 years of age: Lansky score than or equal to 60%.
5. Patients of child-bearing or child-fathering potential must be willing to practice birth control from the time of enrollment on this study and for 4 months after receiving the lymphodepletion regimen.
6. Females of child-bearing potential must have a negative pregnancy test because of the potentially dangerous effects on the fetus.

Patients Exclusion Criteria:

1. Pregnant or lactating women.
2. Severe, uncontrolled active intercurrent infections.
3. HIV, or active HCV and/or HBV infection.
4. Life-expectancy < 6 weeks or rapidly progressive disease that in the evaluation of the investigator would compromise ability to complete study therapy.
5. Hepatic function: inadequate liver function defined as total bilirubin > 4x upper limit of normal (ULN) or transaminase (ALT and AST) > 6x ULN.
6. Renal function: serum creatinine >3x ULN for age.
7. Blood oxygen saturation < 90%.
8. Cardiac function: left ventricular ejection fraction lower than 45% by ECHO.
9. Congestive heart failure, cardiac arrhythmia, psychiatric illness, or social situations that would limit compliance with study requirements or in the opinion of the PI would pose an unacceptable risk to the subject.
10. Presence of active, grade 2-4 acute or chronic Graf versus Host Disease (GvHD) requiring steroid therapy or other immune-suppressive treatment.
11. Relapse occurring before 60 days after alloHSCT.
12. Concurrent or recent prior therapies, before infusion:

    i. systemic steroids (at a dose of ≥ 2 mg/kg prednisone) in the 2 weeks before infusion of CD19-CAR_Lenti_ALLO cells . Recent or recurrent use of inhaled/topical/non-absorbable steroids is not exclusionary.

ii. systemic chemotherapy in the 2 weeks preceding infusion of CD19-CAR_Lenti_ALLO cells .

iii. anti-thymocyte globulin (ATG) or Alemtuzumab (Campath®)in the 8 weeks preceding infusion of CD19-CAR_Lenti_ALLO cells .

iv. immuno-suppressive agentis in the 2 weeks preceding infusion of CD19-CAR_Lenti_ALLO cells

v. radiation therapy must have been completed at least 2 weeks before infusion of CD19-CAR_Lenti_ALLO cells .

vi. other anti-neoplastic investigational agents currently administered or within 30 days prior to infusion of CD19-CAR_Lenti_ALLO cells (i.e, start of protocol therapy).

vii. Exceptions:

1. there is no time restrictions in regards to intrathecal chemotherapy, but there must be a complete recovery from any acute toxic effects from such treatment.
2. subjects receiving steroid therapy at physiologic replacement doses only are allowed provided that there has been no increase for at least 2 weeks to starting apheresis.

Donor Eligibility Criteria

Conventional criteria for the eligibility of allogeneic donors will be adopted for the evaluation of cell donors, before apheresis, as required by law.

Ages: 1 Year to 35 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 24 (Estimated)
Dates: Start 2024-04-28 (Actual); Primary Completion 2026-06-30 (Estimated); Study Completion 2041-06-01 (Estimated)

PRIMARY OUTCOMES:
Safety and establishment of Dose limited Toxicity (DLT) of the infusion of CD19-CAR_Lenti_ALLO cells in pediatric and young adults patients affected by relapsed/refractory BCP-ALL in each dose level | 28 days
  DLT is defined as any of the following events: (1) Grade III-IV GvHD refractory to first and second line treatment and chronic GvHD refractory to first and second-ine treatment; (2) any grade 4 non-hematologic toxicity; (3) grade 4 reactions realted to anti-alloCART infusion; (4) death related to alloCART infusion. The Maximum Tolerated Dose/Recommended Dose (MTD/RD) of CD19-CAR_Lenti_ALLO to be evaluated for efficacy in the phase II extension will be defined as the highest dose level at which <33% of patients (no more than 1 out of 6) experience DLT.

SECONDARY OUTCOMES:
To estimate the rate of occurrence of acute GvHD | 1 year
  The occurrence of acute GvHD will be recorded for every patient
To estimate the severity of acute GvHD (according to the MAGIC criteria) | 1 year
  The severity of acute GvHD will be recorded for every patient
To estimate the rate of occurrence of chronic GvHD | 1 year
  The occurrence of chronic GvHD will be recorded for every patient
To estimate the severity of chronic GvHD (according to the NIH 2014 criteria) | 1 year
  The severity of chronic GvHD will be recorded for every patient
To confirm the safety of the approach at the MTD/RD dose | 28 days
  Toxicity of CD19-CAR_Lenti_ALLO cells will be recorded for every patient
Complete Response (CR) or Complete Response with incomplete blood count recovery (CRi) and MRD negativity achievement. | 28 days
  To evaluate the proportion of patients achieving CR o CR with incomplete blood count recovery (CRi) and MRD negativity by either flow-cytometry or qPCR at day 28 (defined as a value < 1x10^-4)
Probability of CR with MRD negativity achievement according to disease burden at time of enrollment. | 28 days
  To estimate the probability of obtaining CR with MRD negativity stratified according to the disease at time of enrollment (high disease burden being defined as > 5% bone marrow lymphoblasts, any peripheral blood lymphoblasts, Central Nervous System (CNS) 3 status, or non-CNS Extra-Medullary (EM) site of disease.
To assess Overll Survival (OS) in the whole populations of patients. | 1 year
  Overall survival of every patient will be evaluated during follow-up

CONTACTS AND LOCATIONS:
Overall Officials: Franco Locatelli, MD, PhD, Principal Investigator — Director Department of Hematology/Oncology and Cell and Gene Therapy
Locations (1):
- Ospedale Pediatrico Bambino Gesù, Rome, Italy, Italy